

# Clinical Study Protocol CCP-020 (Diacerein 1%) Topical Ointment Sponsor Protocol No. CCP-020-105 TKL Study No. PB710217

# A 6-Week, Randomized Study to Evaluate the Potential of CCP-020 (Diacerein 1%) Topical Ointment to Induce a Photoallergic Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test Design

Author:

Document type: Clinical Study Protocol

Development Phase: 1

Document Date: 25-October-2017

Document Status Final v1.0

Number of Pages: 43

Property of Castle Creek Pharmaceuticals, LLC.

Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Castle Creek Pharmaceuticals, LLC.


**Synopsis** 

Study Title: A 6-Week, Randomized Study to Evaluate the Potential of CCP-020 (Diacerein 1%)

Topical Ointment to Induce a Photoallergic Skin Reaction in Healthy Subjects, Using

a Controlled Photopatch Test Design

TKL Study Number: PB710217

**Sponsor Protocol Number:** CCP-020-105

**Sponsor:** Castle Creek Pharmaceuticals, LLC

**Development Phase:** 1

Study Objectives:

To determine the potential of CCP-020 (Diacerein 1%) Topical Ointment to induce a

photoallergic skin reaction using a controlled photopatch testing procedure.

Study Design: During the 3-week Induction Phase, CCP-020 (Diacerein 1%) Topical Ointment and

vehicle ointment, will each be applied 2 times per week (Monday and Thursday) to 2 sites on the infrascapular area of the back under fully occlusive patch conditions for approximately 24 hours (±4 hours). Minimal erythema dose (MED) irradiation will also be performed for each subject on Day 1. After patch removal, all application sites will be evaluated and one application site of each study product will be irradiated with 2 times the subject's MED using the full Xenon lamp spectrum. All sites will be evaluated at approximately 48 hours later when irradiated on Tuesdays and 72 hours later when irradiated on Fridays. An additional application of study product may be applied on the Monday of rest week 4 if the subject misses an irradiation session during the induction phase of the study. At Challenge, CCP-020 (Diacerein 1%) Topical Ointment and vehicle ointment will each be applied once to 2 naive sites on the infrascapular area of the back under fully occlusive patch conditions for approximately 24 hours (±4 hours). After patch removal, all application sites will be evaluated and one site of each test product will be irradiated with 6 J/cm2 of Ultraviolet A (UVA) followed by 0.5 times the subject's MED of UVA/Ultraviolet B (UVB). An additional untreated site will also be irradiated at Challenge and will serve as an untreated control. Each site, including the untreated control site, will be evaluated again at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) following irradiation. A Rechallenge will be performed if a cutaneous response observed during the Challenge Phase indicates possible

photosensitization or at the discretion of the Investigator.

Planned Sample Size: 50 evaluable subjects

**Study Population:** Healthy adult male and female volunteer subjects

**Investigational Products:** CCP-020 (Diacerein 1%) Topical Ointment

Vehicle Ointment

**Control:** An untreated irradiated non-occlusive (open) control site.

**Efficacy Evaluation** 

Criteria:

Not applicable


Safety Evaluation Criteria:

The safety endpoints for this study are irritation responses during the Induction Phase, positive responses at Challenge (i.e., reactions indicative of a sensitization response) and adverse events. All local and systemic adverse events (AEs) observed by or reported to the Investigator will be evaluated. The intensity, duration, and causal relationship to the study products are to be rated for all AEs.

**Statistical Methods:** 

The focus of the statistical analysis will be the comparison with controls of the photoallergic response to the study products. The diagnosis of photosensitization response will be made by the Investigator based on review of the observed skin responses after Challenge.

Mean numerical equivalent scores, including all scores assigned during Induction, will be analyzed with analysis of variance (ANOVA) with factors subject and treatment. All pairwise treatment comparisons will be performed. Pairs to be compared are: each test sample irradiated versus non-irradiated and all pairwise comparisons on each side.

Number of Study Centers:

Single Center

**Planned Date of Study** 

December 2017 – February 2018

Signature page

**Product names:** 

CCP-020 (Diacerein 1%) Topical Ointment

**Vehicle Ointment** 

**TKL Study number:** 

PB710217

Sponsor protocol number: CCP-020-105

The signatures of the following representatives constitute their approval of this protocol and provide the necessary assurances that this study will be conducted according to all stipulations stated in the protocol, including all statements as to confidentiality. It is also agreed that the study will not be initiated without the approval of an appropriate Institutional Review Board.

## Approved by the following:




# Signature page for the Principal Investigator

**Product names:** 

CCP-020 (Diacerein 1%) Topical Ointment

**Vehicle Ointment** 

TKL Study number:

PB710217

Sponsor protocol number: CCP-020-105

I have read this protocol and agree to conduct this study in accordance with all stipulations of the protocol and in accordance with the Declaration of Helsinki.





# **Table of Contents**

| Synopsis | | 2 |
|------------|----------------------------------------------|----|
| Signature | e page | 4 |
| Signature | e page for the Principal Investigator | 5 |
| Investiga | tors and study administrative structure. | 6 |
| Table of | Contents | 8 |
| List of Ta | ables | 11 |
| List of A | bbreviations | 12 |
| 1. | INTRODUCTION | 13 |
| 1.1. | Background Information | 13 |
| 2. | STUDY OBJECTIVES | 14 |
| 3. | INVESTIGATIONAL PLAN | 15 |
| 3.1. | Study Design | 15 |
| 3.2. | Discussion of Design | 16 |
| 3.3. | Study Population | 16 |
| 3.3.1. | Subject Population | 16 |
| 3.3.2. | Inclusion and Exclusion Criteria | 16 |
| 3.3.3. | Interruption or Discontinuation of Treatment | 18 |
| 3.3.4. | Withdrawals | 19 |
| 3.4. | Treatments | 19 |
| 3.4.1. | Investigational Products and Control. | 19 |
| 3.4.2. | Description of Investigational Products | 21 |
| 3.4.3. | Description of Patch Conditions | 21 |
| 3.4.4. | Packaging/Labeling | 21 |
| 3.4.5. | Assignment to Treatment | 21 |
| 3.4.5.1. | Randomization | 21 |
| 3.4.5.2. | Blinding | 22 |
| 3.4.6. | Prior and Concomitant Therapy | 22 |
| 3.4.7. | Treatment Compliance. | 23 |
| 3.5. | Visit Schedule and Assessments | 23 |
| 3.5.1. | Study Procedures and Visit Schedule | 23 |

| 3.5.2. | Visit Schedule | 26 |
|---|---|---|
| 3.5.3. | Definition of Minimal Erythemal Dose | 28 |
| 3.5.4. | Light source | 28 |
| 3.5.5. | Background information | 28 |
| 3.5.6. | Efficacy Assessments | 28 |
| 3.5.7. | Safety Assessments | 28 |
| 3.5.7.1. | Patch Test Site Evaluations | 28 |
| 3.6. | Adverse Events | 30 |
| 3.6.1. | Method of Determining Adverse Events | 30 |
| 3.6.2. | Adverse Event Definitions | 30 |
| 3.6.2.1. | Adverse Events | 30 |
| 3.6.2.2. | Serious Adverse Events | 31 |
| 3.6.2.3. | Severity of Adverse Events | 32 |
| 3.6.2.4. | Relationship of Adverse Events to Study Treatments | 32 |
| 3.6.3. | Reporting Adverse Events | 32 |
| 3.6.4. | Adverse Event Follow-up | 33 |
| 3.6.5. | Pregnancy reporting | 33 |
| 3.6.6. | Expected Adverse Events | 33 |
| 3.7. | Instructions for Rapid Notification of Serious Adverse Events | 33 |
| 3.7.1. | Contact person and number | 33 |
| 3.7.2. | Reporting Responsibility | 34 |
| 3.7.3. | Reporting procedures | 34 |
| 3.8. | Appropriateness of Safety Measurements | 34 |
| 4. | STATISTICAL METHODS | 35 |
| 4.1. | General Considerations for Data Analysis | 35 |
| 4.2. | Sample Size and Power Considerations | 35 |
| 4.3. | Subject Populations for Analysis | 35 |
| 4.3.1. | Background and Demographic Characteristics | 35 |
| 4.3.2. | Study Product/Visit Compliance | 35 |
| 4.4. | Prior and Concomitant Medications | 36 |
| 4.5. | Efficacy Evaluation | 36 |
| 4.6. | Safety Evaluation | 36 |

| 4.6.1. | Assessment of Responses | 36 |
|--------|------------------------------------------|----|
| 4.6.2. | Photosensitivity | 36 |
| 4.6.3. | Adverse Events | 36 |
| 4.7. | Other topics | 36 |
| 4.8. | Interim analyses | 37 |
| 4.9. | Special Methods | 37 |
| 5. | ADMINISTRATIVE PROCEDURES | 38 |
| 5.1. | Ethics and Good Clinical Practice | 38 |
| 5.2. | Institutional Review Board | 38 |
| 5.3. | Informed consent | 38 |
| 5.4. | Declaration of Helsinki | 39 |
| 5.5. | Changes in Planned Study Conduct | 39 |
| 5.5.1. | Protocol amendments | 39 |
| 5.5.2. | Other changes in study conduct | 39 |
| 5.5.3. | Termination or suspension of study | 39 |
| 5.6. | Data handling and record keeping | 40 |
| 5.6.1. | Recording of data | 40 |
| 5.6.2. | Retention of documents | 40 |
| 5.7. | Product handling and accountability | 40 |
| 5.8. | Quality control and quality assurance | 41 |
| 5.8.1. | Monitoring procedures | 41 |
| 5.8.2. | Auditing procedures | 41 |
| 5.9. | Confidentiality and publication policies | 41 |
| 5.9.1. | Disclosure and confidentiality | 41 |
| 5.9.2. | Communication and publication of results | 42 |
| 6 | REFERENCES | 43 |

## Confidential


# **List of Tables**

| Table 1: | Fitzpatrick Skin Types | 24 |
|----------|----------------------------------|----|
| Table 2: | Visit Schedule and Assessments | 27 |
| Table 3: | Response Scores | 29 |
| Table 4: | Notations | 29 |
| Table 5: | Relationship of AE to Study Drug | 32 |

## **List of Abbreviations**

AE Adverse Event

ANOVA Analysis of Variance

CFR Code of Federal Regulations

CRF Case Report Form
DMP Data Management Plan

EBS Epidermolysis bullosa simplex

EOS End of Study

FDA Food and Drug Administration

GCP Good Clinical Practice

GMP Good Manufacturing Practice
IB Investigational Brochure

ICH International Conference on Harmonisation

ICF Informed Consent Form
IP Investigational Product
IRB Institutional Review Board
MED Minimal Erythemal Dose

MedDRA Medical Dictionary for Regulatory Activities

NF National Formulary

NSAIDs Non-Steroidal Anti-Inflammatory Drugs

OA Osteoarthritis
OTC Over-the-counter
PI Principal Investigator
PMD Primary Medical Doctor
SAE Serious adverse event
SAP Statistical Analysis Plan

SOPs Standard Operating Procedures

TKL TKL Research, Inc.
UPT Urine pregnancy test

USP United States Pharmacopeia

UV Ultraviolet
UVA Ultraviolet A
UVB Ultraviolet B

## 1. INTRODUCTION

This study evaluates the potential of CCP-020 (Diacerein 1%) Topical Ointment to induce a photoallergic skin reaction using a controlled photopatch test design. Because CCP-020 (Diacerein 1%) Topical Ointment is formulated for topical use, it is necessary to determine the potential of this product to cause a photoallergic reaction after application to the skin.

The study will be conducted in compliance with Food and Drug Administration (FDA) regulations, the ethical principles of the Declaration of Helsinki concerning medical research in humans (Recommendations Guiding Physicians in Biomedical Research Involving Human Subjects, Helsinki 1964 and amendments 2013), the International Conference on Harmonization (ICH) – Good Clinical Practice (GCP) Guidelines as currently amended, and all applicable standard operating procedures (SOPs) of TKL Research, Inc. (TKL).

## 1.1. Background Information

CCP-020 (previously developed as AC-203) is a topical ointment containing diacerein (4,5-bis[acetyloxy]-9,10-dihydro-9,10-dioxo-2-anthracene carboxylic acid; also known as diacetylrhein), a highly purified anthraquinone derivative, and is being developed by Castle Creek Pharmaceuticals for the treatment of epidermolysis bullosa simplex (EBS). The capsule formulation of diacerein, intended for oral use and systemic absorption, was initially approved for use in osteoarthritis (OA) in France in 1992 (as Artodar®, ART50®, or Zondar®). Since then, it has received marketing authorization in over 30 countries in Europe, South America, and Asia. It is classified as a Symptomatic Slow-Acting Drug in OA. Following oral administration of the capsule formulation, diacerein is rapidly metabolized to the deacetylated active metabolite, rhein. Similarly, diacerein in the topical formulation is hydrolyzed to rhein in the epidermis and the dermis following administration. Diacerein and rhein have been shown to inhibit the in vitro and in vivo production and activity of interleukin (IL)-1 $\beta$  and other proinflammatory cytokines. It has a novel mode of action that differentiates it from non-steroidal anti-inflammatory drugs (NSAIDs) and other conventional forms of drug therapy.

For the development of CCP-020, a total of 10 animal studies have been conducted with CCP-020 ointment 1%, including one skin penetration study, three acute dermal toxicity studies, one phototoxicity study, three pharmacokinetic studies, and two sub-chronic juvenile toxicity studies. CCP-020 was well-tolerated in these studies and no untoward adverse effects (AEs) were noted. To date, two clinical studies of CCP-020 have been completed in patients with epidermolysis bullosa simplex (EBS). These include a Phase one pilot study in five patients and a Phase 2, multiple-site study in 17 patients in Europe. The Phase 2 study demonstrated CCP-020 was well-tolerated and no treatment-related AEs were reported. The Investigator's Brochure should be consulted for summaries of the results of these studies.<sup>1</sup>

This Phase 1 study will assess the photoallergic potential of CCP-020 (Diacerein 1%) topical ointment.


# 2. STUDY OBJECTIVES

The objective of this study is to determine the photoallergic potential of CCP-020 (Diacerein 1%) topical ointment when topical application to skin is followed by light exposure.

In addition, safety will be assessed by evaluation of any adverse events (AEs) reported during the study.

## 3. INVESTIGATIONAL PLAN

# 3.1. Study Design

This will be a randomized, double-blind, single-center, vehicle-controlled, within-subject comparison study of the study products, CCP-020 (Diacerein 1%) topical ointment, vehicle ointment, and an untreated irradiated non-occluded (open) control site. A total of 4 application sites (2 cm x 2 cm each) will be marked on the subject's back and distributed so that 2 sites are on each side of the back. One side of the back will be designated for irradiation after approximately 24 hours (±4 hours) of study product application and the other side will remain non-irradiated. An additional site will be marked on the "irradiated side" of the back. The site will receive no study product, but will be irradiated at Challenge to serve as an untreated irradiated non-occluded control.

A defined area (approximately 50 cm<sup>2</sup>) on the infrascapular region of each subject's back will be irradiated to determine the minimal erythemal dose (MED) of ultraviolet (UV) light.

During the 3-week Induction Phase, 0.2 mL of each study product will be applied to 2 sites twice each week (Monday and Thursday) for approximately 24 hours (±4 hours) under occlusive patch conditions (6 applications). After patch removal, all application sites will be evaluated and one application site of each study product will be irradiated with 2 times the subject's MED using the full Xenon lamp spectrum. The sites will be evaluated by a trained evaluator. All sites will be reevaluated post irradiation, at approximately 48 hours later when irradiated on Tuesdays and at approximately 72 hours later when irradiated on Fridays except when irradiated on the last Friday of the Induction Phase or if a subject is taking a missed visit during induction, the sites will not be evaluated. These procedures will be performed each week for 3 weeks of the Induction Phase. Dermal reactions at the application sites will be evaluated using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation (see Table 3 and Table 4).

At the end of the Induction Phase, the subjects will enter a Rest Period of 10-17 days and then a Challenge Phase. One application/irradiation session may be missed during the Induction Phase. It must be made-up during Week 4. An additional application of study product may be applied on the Monday of rest week 4 if the subject had missed an irradiation session during the induction phase of the study. In either case, no evaluation will be required following irradiation.

At Challenge, each study product will be applied in an amount of 0.2 mL to 2 naive sites once for approximately 24 hours (±4 hours) under occlusive patches. After 24 hours (±4 hour) of product application, all sites will be evaluated and one application site of each product and the additional untreated control site will be irradiated. The sites will be examined for dermal reactions at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) post-irradiation. A Rechallenge will be performed if a cutaneous response observed during the Challenge Phase indicates possible photosensitization or at the discretion of the Investigator.

The safety endpoints for this study are irritation responses during the Induction Phase, positive responses at Challenge (i.e., reactions indicative of a sensitization response) and adverse events

# 3.2. Discussion of Design

Results are interpreted according to working criteria which are based upon published works, as well as the clinical experience of TKL Research, Inc. These working criteria are periodically reviewed and amended subject to new information that becomes available.

This photoallergy study is designed to detect the ability of the CCP-020 (Diacerein 1%) topical ointment and vehicle ointment to cause photoallergic skin reactions when exposed to sunlight. Each subject is to receive applications of the CCP-020 (Diacerein 1%) topical ointment and the vehicle ointment product to 2 separate sites. One will be irradiated and one will remain non-irradiated. An untreated non-occluded control site will also be irradiated at Challenge. This design provides built-in controls for the test product CCP-020 (Diacerein 1%) topical ointment under both irradiated and non-irradiated conditions.

# 3.3. Study Population

## 3.3.1. Subject Population

A sufficient number of subjects will be enrolled in order to provide 50 completed subjects evaluable for analysis; an individual subject will be allowed to participate in the study one time only.

A rationale for the choice of sample size is provided in Section 4.2 of this protocol.

#### 3.3.2. Inclusion and Exclusion Criteria

#### **Inclusion Criteria**

A subject will be considered eligible for participation in the study if all of the following inclusion criteria are satisfied prior to randomization:

- 1. Is a healthy male or female (to be confirmed by medical history);
- 2. Is 18 years of age or older;
- 3. In the case of a female of childbearing potential, is using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy, tubal ligation). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
- 4. In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) at Day 1 and are willing to submit to a UPT at the end of study (EOS);
- 5. Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;

- 6. Has uniformly-colored skin on the lower thoracic area of the back which will allow discernment of erythema, and has Fitzpatrick Skin Types I, II, or III (see Table 1);
- 7. Complete a medical screening procedure; and
- 8. Read, understand, and sign an informed consent.

#### **Exclusion criteria**

A subject who has any of the following will be excluded from the study:

- 1. Has a history of photosensitivity or photoallergy;
- 2. Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
- 3. Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
- 4. Is not willing to refrain from using systemic/topical anti-inflammatory analysis such as aspirin (81 mg daily aspirin will be allowed), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
- 5. Are taking medication known to cause phototoxic reactions (eg, tetracyclines, thiazides, nonsteroidal anti-inflammatory drugs [NSAIDS]);
- 6. Is using medication which, in the opinion of the Investigator, will interfere with the study results (e.g. anti-inflammatory medications, antipsychotics, anticonvulsants with potential pain relief effects, immunomodulatory medications, and others);
- 7. Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
- 8. Has psoriasis and/or active atopic dermatitis/eczema;
- 9. Has a known sensitivity or allergy to constituents of the materials being evaluated including diacerein, mineral oil, petrolatum, cetyl alcohol, D&C Yellow #10 and/or ethyl paraben;
- 10. Is a female who is pregnant, plans to become pregnant during the study, or is breast feeding a child;
- 11. Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
- 12. Has received treatment for any type of internal cancer within 5 years prior to study entry;
- 13. Has a history of, or are currently being treated for skin cancer and/or hepatitis;
- 14. Has a history of, or is currently being treated for diabetes;
- 15. Has any condition that might compromise study results;
- 16. Currently or expect to sunbathe or use tanning salons during the study;

- 17. Has a history of adverse response (eg, blistering, sun poisoning) to ultraviolet (UV) sun lamps/sunlight exposure;
- 18. Is currently participating in any clinical testing;
- 19. Has any known sensitivity to adhesives; and/or
- 20. Has received any investigational drug(s) within 4 weeks prior to study entry.

## 3.3.3. Interruption or Discontinuation of Treatment

A reaction of at least moderate erythema (2) accompanied with mild, but definite edema (1) to a study product observed after the first patch application/irradiation sequences of the Induction Phase may indicate the subject to be pre-sensitized, and may cause the discontinuation of the subject from the study.

After the second reading of the Induction Phase, either of the following conditions will require the study product be applied to a naive patch site under semi-occlusive patch conditions:

- Reaction of >50% "p" or "p" with no erythema, minimal/doubtful erythema, or definite erythema; or "D" (see Tables 3 and 4);
- Any reaction of definite erythema with definite edema.

Study product may not be relocated more than twice.

The 3 weeks of continuous patch contact during the Induction Phase frequently results in tape-related irritation that is exacerbated by warm weather, but which occurs among some individuals irrespective of the season. Tape-related irritation will not be graded as a photosensitivity response at the patch site, but will be noted separately on the CRF. Severe tape-related irritation will necessitate a change in the application site. As above, the application site will only be changed twice and then the subject must be discontinued.

One application/irradiation session may be missed during the Induction Phase. It must be made-up during Week 4. In this case, no evaluation will be required following irradiation. Only one missed patch application for study product is allowed. A subject must be discontinued and considered not complete if more than one application is missed.

In accordance with legal requirements and ICH-GCP guidelines, every subject or his/her legal representative has the right to refuse further participation in the study at any time and without providing reasons (see also Section 5.3). A subject's participation is to be terminated immediately upon his/her request. The Investigator should seek to obtain the reason and record this on the case report form (CRF).

If at the time of refusal a study product has already been administered, the subject should be advised on follow-up safety investigations. If a subject withdraws from the study, all efforts will be made to complete a final evaluation if possible. Subjects discontinued for having experienced an AE will be followed until the AE is resolved, a reasonable explanation is provided for the event, or the subject is referred to his/her own primary medical doctor (PMD). The specific AE in question will be recorded on the appropriate CRF.

If a subject develops a serious adverse event (SAE), his/her termination from the study will be considered by the Investigator. Similarly, if the subject develops conditions over the course of

the study which would have excluded his/her entry in the study according to the safety-related medical exclusion criteria, he/she must be withdrawn immediately.

The subject may be withdrawn from the study at any time at the discretion of the Investigator for medical reasons and/or due to non-adherence to the treatment scheme and other duties stipulated in the study protocol. The reasons are to be documented on the CRF.

In addition, the Sponsor retains the right to end the study at any time if the study cannot be carried out as agreed upon in the protocol. In case of premature termination or suspension of the study, the Sponsor's study manager will promptly inform the Investigator/institutions and regulatory authorities of the termination or suspension and the reason for that. It is the responsibility of the Principal Investigator (PI) to notify the Institutional Review Board (IRB) in the case of premature termination/suspension.

#### 3.3.4. Withdrawals

The following medical and other reasons justify a premature termination (by subject or Investigator) of any of the study IPs.

- Adverse Event/Serious Adverse Event
- Death
- Protocol Violation (e.g. non-compliance)
- Investigator Judgment
- Pregnancy
- Lost to Follow-up
- Withdrawal by Subject
- Study Terminated by Sponsor
- Other

If a subject withdraws from the study, all efforts will be made to complete a final evaluation, if possible. Subjects discontinued for having experienced an AE will be followed until the AE is resolved, a reasonable explanation is provided for the event, or the subject is referred to his/her own primary medical doctor (PMD). The specific AE in question will be recorded on the appropriate CRF.

#### 3.4. Treatments

## 3.4.1. Investigational Products and Control

## **Investigational Product(s):**

#### CCP-020 (Diacerein 1%) Topical Ointment

CCP-020 is a topical ointment, 1% (w/w). All excipients used in the topical formulation meet United States Pharmacopeia (USP)/ National Formulary (NF) criteria and are commonly used in

ointment formulations. CCP-020 (Diacerein 1%) topical ointment is packaged in aluminum tubes, at 25 g/tube.



CCP-020 topical ointment and vehicle ointment should be stored at room temperature (15°C/59°F to 30°C/86°F). The PI will be responsible for the suitable storage of the IPs in compliance with the storage instructions and must restrict access to the investigative personnel

Lot numbers will be given in the clinical study report.

Manufacturer:



## Control

An untreated irradiated non-occlusive (open) 2 cm x 2 cm site will serve as a control.

## 3.4.2. Description of Investigational Products

CCP-020 (Diacerein 1%) topical ointment and vehicle ointment will be supplied in aluminum tubes for the clinical study. CCP-020 (Diacerein 1%) topical ointment and vehicle ointment were manufactured and packaged in accordance with good manufacturing practice (GMP).

## 3.4.3. Description of Patch Conditions

Material evaluated under occlusive patch conditions is applied to a 2 cm x 2 cm Webril® pad attached to a non-porous, plastic film adhesive bandage (medical tape). The patch is secured with hypoallergenic tape (Micropore), as needed.

## 3.4.4. Packaging/Labeling

The study medication tube label will show at least the following:

- Protocol number
- Storage conditions
- Instructions for use
- Expiration date
- Sponsor information
- Investigational drug warning
- Space to enter lot number.

A full product description can be found in the Investigator's Brochure (IB).<sup>1</sup>

All study IPs should be stored at room temperature (15°C/59°F to 30°C/86°F).

## 3.4.5. Assignment to Treatment

#### 3.4.5.1. Randomization

Each subject who signs an informed consent form (ICF) will be assigned a screening number. If the subject meets all of the inclusion and none of the exclusion criteria, and successfully completes the screening procedures, they will be enrolled in the study. Upon enrollment, each subject will be assigned a unique subject number and receive a randomization code, indicating application placement of the study materials. Each subject in this study will serve as his or her own control. All subjects will receive the IPs and control products at adjacent application sites, i.e. study product placement on the left side of the back will be the same as on the right side of the back.

CCP-020 (Diacerein 1%) topical ointment and vehicle ointment will be assigned in a randomized sequence to the test sites. The same study material will be applied to the same test site throughout the study.

## **3.4.5.2.** Blinding

CCP-020 (Diacerein 1%) topical ointment, vehicle ointment, and control will not be blinded to investigative personnel involved in the preparation/application and removal of treatments.

Investigative personnel who are involved in the preparation/application and removal of the treatments will be unblinded and will not perform the evaluation of skin responses. The subjects and the trained evaluator who will be evaluating skin responses will be blinded to IPs and the treatment allocation; however, because of the demarcations/skin coloration remaining on the skin following patch removal, complete blinding of the evaluators cannot be completely assured.

Investigative personnel who are blinded, including the Investigator and trained evaluator involved in the evaluation of responses, will remain blinded during the course of the study until Database Lock and finalization of the Statistical Analysis Plan (SAP).

In the event of an emergency, if possible, the Investigator or designee will contact the Sponsor with notification of the intent to unblind the treatment codes prior to the actual unblinding. If it is not possible to notify the Sponsor prior to the unblinding, the Investigator or designee will contact the Sponsor immediately following the unblinding procedure and follow with a written notification to document the exact manner in which the code was broken and the justification for the unblinding. The Investigator will communicate the treatment identification to only the investigative personnel who require the information to manage the emergency. Unblinding will happen on site at TKL.

## 3.4.6. Prior and Concomitant Therapy

All medications, including over the counter (OTC) drugs and vitamins, taken within 28 days prior to the start of the study will be recorded at Screening. Thereafter, a record of all medications taken during the course of the study will be made. Information regarding the total daily dose, route of administration, start and discontinuation dates, and indication are to be captured on the subject's CRF.

The following prohibitions will apply for the duration of the study:

- There will be no use of systemic/topical anti-inflammatory analgesics which in the opinion of the investigative personnel will interfere with the study results, including anti-inflammatory medications such as aspirin (81 mg aspirin will be allowed at the discretion of the Investigator), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
- Use of sunbeds or sunlamps or deliberate exposure of the test sites to natural sunlight or to other sources of UV light;
- Participation in any other clinical study;
- Soaking of test areas; and/or
- Application of any product to the test areas.

The use of or change in the dose of any and all concomitant medication, either prescription or OTC, during the study will be recorded. The reason for use or change of dose of a concomitant therapy may need to be reported as an AE. Therapies (medication and non-medication therapies)

not restricted by the protocol may be used. Non-prohibited chronic therapies being used at Baseline may be continued.

All topical or systemic medication listed in the exclusion criteria are prohibited during this study. See the IB for information about possible drug-drug interactions.<sup>1</sup>

#### 3.4.7. Treatment Compliance

All patches will be applied and removed by investigative personnel. Whereas bathing will be allowed (low tub bath/frontal showers), the patched areas are not to be soaked and are to be kept as dry as possible, per the instructions to be given to each subject. Subjects will be instructed to contact the Investigator before starting any medication, including OTC remedies. In the case of an emergency treatment, the Investigator must be informed as soon as possible. A trained, experienced evaluator will assess study compliance.

Records of patch applications and visit schedule compliance will be recorded on the subjects' CRFs.

## 3.5. Visit Schedule and Assessments

## 3.5.1. Study Procedures and Visit Schedule

## **Screening**

At Screening, the subjects will receive any necessary written and verbal information, and the informed consent of each subject will be obtained. Demographic data (including Fitzpatrick skin type) will be recorded, a medical history will be taken, and previous and concomitant medications will be reviewed. Eligibility will be determined by review of the inclusion/exclusion criteria.

- Any written and verbal information
- Informed consent
- Demographics
- Previous/concomitant medication
- Review of inclusion and exclusion criteria
- Medical history (including lifestyle and habits)
- Evaluation of application site area

| Table 1: | Fitzpatrick Skin Types |
|----------|----------------------------------------------|
| I | Always burns easily, never tans |
| II | Always burns easily, tans minimally |
| III | Burns moderately, tans gradually |
| IV | Burns minimally, always tans well |
| V | Rarely burns, tans very well |
| VI | Never burns, deeply pigmented <sup>3,4</sup> |

## Day 1

On Day 1, all subjects will be questioned regarding the entry criteria and female subjects of childbearing potential will undergo a UPT. If the subject fulfills all the inclusion and none of the exclusion criteria, he/she will be allowed participation in the study. Upon enrollment, each subject will be assigned a unique subject number and receive a randomization code, indicating application placement of the study products.

A baseline evaluation of the patch sites will be performed immediately prior to application of the patches to ensure that no conditions, markings, or coloration of the skin will interfere with interpretation of the study results.

A total of 4 application sites (2 cm x 2 cm each) will be marked on each subject's back, placing 2 sites on opposite sides of the back. The distance between the patches will be no less than one centimeter. The numbering of the test sites will remain the same throughout the study. The sites will be marked with an indelible, surgical marker.

## Minimal Erythema Dose (MED) Determination

On Day 1, subjects will have an area of skin on their back, approximately 50 cm<sup>2</sup>, divided into 6 equal sites marked with a surgical marker. Each of the sites will be irradiated with full spectrum UV light, with each exposure differing from the next by a factor of 1.25 (ie, each irradiated site will be exposed to a 25% greater dose of UV irradiation than the previous site).<sup>2</sup>

The areas involved in MED determination will be different from the study product application sites. Evaluation of the exposed sites will be performed on Day 2.


#### Induction

The Induction Phase consists of a series of 4 patch applications of the study products and subsequent irradiation and evaluations of the patch test sites over a 3-week Induction Phase.

Under occluded conditions, 0.2 mL of each study product, CCP-020 (Diacerein 1%) topical ointment and vehicle ointment will be applied to two Webril® pads. The patches will be secured with nonporous plastic film adhesive bandage (Blenderm tape) and hypoallergenic paper tape (3M Micropore<sup>TM</sup>), as needed. The patches will then be applied to their assigned sites on each side of the back for 24 hours (±4 hours). This process will be repeated twice each week (Mondays and Thursdays) during the 3-week Induction Phase. The same study product will be applied to the same test site throughout the Induction Phase.

Application sites will be evaluated immediately prior to study product application.

After 24 hours (±4 hours) of study product application (eg, Tuesday and Friday), all patches will be removed. The sites will be evaluated using the scoring system detailed in Section 3.5.7.1. One side of the back will be assigned for irradiation and the other will remain non-irradiated, ie, only one application site of each study product will receive irradiation. On all Tuesdays and Fridays, the sites designated for irradiation will be irradiated with 2 times the subject's MED using the full Xenon lamp spectrum.

Adverse events and concomitant medications will be reviewed at each visit and recorded as applicable.

One application/irradiation session may be missed during the Induction Phase. It must be made-up during Week 4. An additional application of study product may be applied on the Monday of rest week 4 if the subject misses an irradiation session during the Induction Phase of the study. No evaluation will be required following the final irradiation during the challenge period.

## Rest Period (Weeks 4 and 5)

During the Rest Period of approximately 10-17 days, subjects will not receive any application of study materials. An additional application of study product may be applied on the Monday of rest week 4 if the subject misses an irradiation session during the Induction Phase of the study.

#### Challenge (Week 6)

On Day 1 of the Challenge Phase, subjects who have completed the Induction Phase and the Rest Period will have study product applications to naive sites in the same manner as applied during the Induction. A baseline evaluation of the naïve sites will be performed immediately prior to application of the patches to ensure that no conditions, markings, or coloration of the skin will interfere with interpretation of the study results. As in the Induction Phase, 0.2 mL of CCP-020 (Diacerein 1%) topical ointment and vehicle ointment will each be applied to 2 naive sites for approximately 24 hours (±4 hours) under occlusive patch conditions. The clinical staff will then remove the patches and a trained evaluator will evaluate the test sites. There will be a main evaluator for the study; a backup evaluator will also be assigned in the event that an emergency occurs and the main evaluator is unable to attend the study visit. The designated sites and an additional untreated control site will be irradiated with 6 J/cm<sup>2</sup> of UVA (320-400 nm) followed by 0.5 times the MED of UVA/UVB (full-spectrum) irradiation, obtained by using a filtered light

source (see Section 3.5.4). Each site will be evaluated again at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) post irradiation.

Adverse events and concomitant medications will be reviewed at each visit and recorded as applicable. A UPT will be performed for female subjects of childbearing potential at the last study visit.

#### Rechallenge

A Rechallenge should be performed if a cutaneous response observed during the Challenge Phase indicates possible photosensitization or at the discretion of the Investigator. If it is determined by the Investigator that a Rechallenge should be performed, the Rechallenge patches will be applied as soon as Challenge reactions have resolved. Just as in the challenge procedure 0.2 mL of each study product CCP-020 (Diacerein 1%) topical ointment and vehicle ointment, will each be applied to 2 naive sites for approximately 24 hours (±4 hours) using appropriate patches to further discriminate a photosensitization reaction from an irritation reaction. A baseline evaluation of the naïve sites will be performed immediately prior to application of the patches to ensure that no conditions, markings, or coloration of the skin will interfere with interpretation of the study results. Approximately twenty-four (24) hours (±4 hours) after study product application, the clinical staff will remove the patches and a trained evaluator will evaluate the test sites. One site of each product and an additional untreated control site will be irradiated with 6 J/cm<sup>2</sup> of UVA (320-400 nm) followed by 0.5 times the MED of UVB (290-320 nm) irradiation using a filtered light source. All sites (irradiated and non-irradiated) will be graded for dermal reactions at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) following irradiation. Concomitant medications and AEs will also be reviewed.

## **End of Study**

At the EOS, all patches will be removed as described above, and the final evaluations of the test sites will be made.

An EOS examination will be conducted and consist of the following:

- Concomitant medication
- AEs
- UPT in females of childbearing potential

Concomitant medications and AEs will be reviewed and recorded during the whole study. For a detailed listing of scheduled study time points refer to the Visit Schedule and Assessments (Table 2).

## 3.5.2. Visit Schedule

A summary of the visit schedule and assessments is presented in Table 2.

**Table 2:** Visit Schedule and Assessments

| | Screening | Day<br>1 <sup>a</sup><br>(M) | Induction | | | Rest | Challenge<br>(Week 6) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | , | | M<br>8,<br>15 | Tu<br>2,<br>9,<br>16 | Th<br>4,<br>11,<br>18 | F<br>5.<br>12,<br>19 | Week<br>4 & 5 | M | Tu | W | Th | F |
| Informed consent | X | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | |
| Demographic information | X | | | | | | | | | | | |
| Fitzpatrick Skin<br>Typing | X | | | | | | | | | | | |
| UPT | | X | | | | | | | | | | X |
| MED irradiation/evaluation | | Xb | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | |
| Product application | | X | X | | X | | | X | | | | |
| Application site evaluations | | | Xc | X | X | X <sup>d</sup> | | | X | X | X | X |
| Application site irradiation | | | | X | | X <sup>d</sup> | | X | X | | | |
| Make-up evaluation/application | | | | | | | Xe | | | | | |
| Make-up evaluation/<br>irradiation | | | | | | | Xe | | | | | |
| Review of concomitant medications | X | X | X | X | X | X | X <sup>f</sup> | X | X | X | X | X |
| Review of AEs | X | X | X | X | X | X | X <sup>f</sup> | X | X | X | X | X |

- a Screening and the first day of Induction (Day 1) may take place on the same day.
- b MED irradiation on Day 1 and MED evaluation on Day 2.
- c The first Monday (Week 1) of the Induction Phase.
- d Evaluations will not be conducted after irradiation on the last Friday of the Induction Phase. Untreated control site will also be irradiated.
- e Make-up evaluation/application and evaluation/irradiation are performed as necessary (see Section 3.5.1).
- f Concomitant medications and AEs will be reviewed only for subjects who are required to return to the test facility for make-up visits during Rest Period Week 4.

**Note:** The visit schedule may be revised if necessary.

## 3.5.3. Definition of Minimal Erythemal Dose

Minimal erythemal dose (MED) is defined as the length (in time) of light exposure required to produce a minimal erythema reaction 16 - 24 hours after irradiation using a standardized filtered UV light source that emits UVB (290-320 nm) as part of its emission spectrum.<sup>2</sup>

## 3.5.4. Light source

The light source will be a Xenon Arc Solar Simulator (150 W), with UV-reflecting dichroic mirror, UVC-blocking filter, and visible/infrared blocking filter to generate a continuous emission spectrum in the UVA and UVB range (290 to 400 nm).<sup>2</sup> An additional filter is added during irradiation of the application sites to block UVB radiation allowing only UVA irradiation of the sites. The output is measured daily prior to irradiation using a radiometer/photometer.

## 3.5.5. Background information

Date of birth, gender, race, Fitzpatrick skin type (see Table 1), and a significant medical history of each subject will be recorded at Screening.

## 3.5.6. Efficacy Assessments

No efficacy will be assessed in this study.

## 3.5.7. Safety Assessments

## 3.5.7.1. Patch Test Site Evaluations

For both Induction and Challenge Phases, after 24 hours (±2 hour) of product application, all sites will be evaluated and one application site of each product and the additional untreated site will be irradiated. The sites will be examined for dermal reactions at approximately 24 hours (±4 hours), 48 hours (±4 hours), and 72 hours (±4 hours) post-irradiation.

The scores in Table 3 will be used to express the response observed at the time of examination and will be recorded on the subjects' CRFs. The score will be used for statistical analysis. Additional response notations are presented in Table 4.

**Table 3:** Response Scores

| Response | Symbol | Numerical<br>Equivalent Score |
|---|---|---|
| Erythema | | |
| No reaction | - | 0 |
| Mild, but definite erythema | + | 1 |
| Moderate erythema | ++ | 2 |
| Marked/severe erythema | +++ | 3 |
| Edema | | |
| No reaction | - | 0 |
| Mild, but definite edema | ** | 1 |
| Definite edema with erosion/vesiculation | *** | 2 |

**Table 4:** Notations

| Response/Comment | Notation |
|---|---|
| Hyperpigmentation | Hr |
| Hypopigmentation | Но |
| Vesiculation | V |
| Papular response | p |
| Papulovesicular response | pv |
| Damage to epidermis: oozing, crusting, and/or superficial erosions | D |
| Itching | I |
| Spreading of reaction beyond patch study site (ie, reaction where material did not contact skin) | S |
| Follicular irritation with or without pustule formation (folliculitis) | f |
| Subject absent | X |
| Patch dislodged | PD |
| Not patched | NP |
| No reaction | 0 |

The readings will be made under a standardized white light source.

The 3-week period of patch contact during the Induction Phase may result in tape-related irritation in some individuals. Tape related irritation will not be graded as an irritant response at the patch site but will be noted separately on the CRF.

The Investigator will assess the reactions seen during the Challenge Phase and determine whether the subject is photosensitized or not. The following guidelines are generally considered in this assessment. Not all observations of erythema and edema are associated with photosensitivity; only if erythema and edema are observed can a reaction be suspected of being a positive photosensitivity reaction. An increase in the intensity of the reaction over time further

supports an assessment of photosensitivity. If reactions are observed at both the irradiated and non-irradiated study product sites (ie, if contact sensitization may have occurred), the reaction at the irradiated site upon Rechallenge must be at least one grade more intense than at the non-irradiated site for the reaction to be suspected of being a photosensitivity reaction (refer to Section 3.5.7.1 for response scores and notations).

#### 3.6. Adverse Events

## **3.6.1.** Method of Determining Adverse Events

Safety assessments will include recording AEs reported spontaneously by the subject or collected by the Investigator. AEs will be recorded at each visit throughout the study on the appropriate CRF. Every attempt should be made to describe the AE in terms of a diagnosis. If a clear diagnosis has been made, individual signs and symptoms will not be recorded unless they represent atypical or extreme manifestations of the diagnosis, in which case they should be reported as separate events.

Subjects should be asked whether, since the time of the last observation or visit, they had any of the following:

- Experience any changes in well-being;
- Used any new medications;
- Changed medication regimens (both prescription and OTC); and/or
- Were admitted to a hospital or had any accidents.

All questions should be of a general nature and should not suggest symptoms.

When an AE is suspected, all relevant evaluations will be carried out and appropriate treatment provided. Additional follow-up will be done as necessary (Section 3.6.4) and recorded in the subject's source documents, and the results will be provided to the Sponsor.

For AE definitions and reporting requirements refer to Section 3.6.2 and Section 3.6.3.

Note: Any observed response which can be denoted using the irritation criteria summarized in Table 3 and Table 4 will not be considered an AE. Likewise, any tape-related irritation will only be noted as an AE when all patches are discontinued due to tape reaction around all sites (see Section 3.6.6).

#### 3.6.2. Adverse Event Definitions

#### 3.6.2.1. Adverse Events

Information about all local and systemic AEs, whether volunteered by the subject, discovered by Investigator questioning, or detected through other means, will be collected and recorded on the AE CRF and followed as appropriate.

An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product (or cosmetic product), which does not necessarily have a causal relationship with this treatment. An AE can therefore, be any unfavorable and

unintended sign, symptom, or disease temporally associated with the use of a medicinal investigational product, whether or not considered related to the medicinal investigational product.

Adverse Events will be coded using an internationally recognized dictionary (MedDRA).

Medical conditions/diseases present before starting study treatment are considered AEs only if they worsen after starting study treatment (any procedures specified in the protocol). Any AEs occurring before starting study treatment but after signing the ICF are recorded on the Medical History/Current Medical Conditions CRF.

To the extent possible, each AE will also be described by:

- 1. its duration (start and end dates),
- 2. the severity grade (mild, moderate, severe)
- 3. its relationship to the study drug,
- 4. the action(s) taken, and
- 5. as relevant, the outcome.

Note: Any observed response which can be denoted using the irritation criteria summarized in Table 3 and Table 4 will not be considered an AE. Likewise, any tape-related irritation will not be noted as an AE.

#### 3.6.2.2. Serious Adverse Events

A "SAE" is any AE that:

- Results in death;
- Is life-threatening (Note: the term "life-threatening" refers to any AE that, as it occurs, puts the subject at immediate risk of death. It does not refer to an AE that hypothetically might have caused death if it were more severe).
- Results in hospitalization or prolongation of current hospitalization (not including
  hospitalization for a pre-existing condition that has not increased in severity or
  frequency from the subject's underlying medical condition prior to entry into the
  study).
- Is a congenital anomaly/birth defect in the offspring of a subject.
- Is another serious (important medical events) event.
- Results in persistent or significant disability/incapacity.

(Note: Important medical events may not be immediately life-threatening or result in death or hospitalization but may be considered serious when, based on the appropriate medical judgment, they may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home; blood dyscrasias or convulsions that do not result in inpatient hospitalization; or development of drug dependency or drug abuse.)

## 3.6.2.3. Severity of Adverse Events

"Severity" of the AE refers to the extent to which an AE affects the subject's daily activities and differs from "Serious," which is a regulatory classification.

The Investigator is to classify the severity of an AE according to the following definitions:

- **Mild:** The symptom has a negligible effect or no impairing effect on the subject's normal function.
- **Moderate:** The symptom impairs the subject's normal function to some extent.
- **Severe:** The symptom has an obvious, significantly impairing effect on the subject's normal function.

## 3.6.2.4. Relationship of Adverse Events to Study Treatments

The Investigator is to classify the drug relationship of an AE according to the definitions outlined in Table 5.

Table 5: Relationship of AE to Study Drug

| Association | Definition |
|---|---|
| Not related | (1) the existence of a clear alternative explanation (e.g., mechanical bleeding at surgical site) or (2) non-plausibility, e.g., the subject is struck by an automobile or cancer developing a few days after drug administration. |
| Unlikely | There is no medical evidence to suggest that the AE may be related to study drug usage, or there is another more probable medical explanation. |
| Possible | There is medical evidence to suggest that there is a reasonable possibility that the AE may be related to study drug usage. However, other medical explanations cannot be excluded as a possible cause. |
| Probable | There is strong medical evidence to suggest that the AE is related to study drug usage. |
| Definite | A clinical event, including laboratory test abnormality (if applicable), in which there is no uncertainty in its relationship to test drug (e.g., positive Rechallenge). |

## 3.6.3. Reporting Adverse Events

Adverse events that occur from the time of informed consent through completion of the last study visit should be reported.

Every attempt should be made to describe the AE in terms of a diagnosis. If a clear diagnosis has been made, individual signs and symptoms will not be recorded unless they represent atypical or extreme manifestations of the diagnosis, in which case they should be reported as separate events. If a clear diagnosis cannot be established, each sign and symptom must be recorded individually.

Any SAEs occurring in a subject receiving study drug must be reported to the Sponsor within 24 hours of the site being informed of the event, even if the event does not appear to be drug-

related. The report must be made by sending a completed SAE Report form to the Sponsor. Any pertinent follow-up information should be provided in a similar manner. Contact information is provided in Section 3.7.1.

## 3.6.4. Adverse Event Follow-up

Any ongoing AE at the time of study completion or withdrawal will be followed until the AE is resolved or the subject is referred to his/her own PMD. The Investigator and the Sponsor will decide if longer follow-up is appropriate on a case-by-case basis. Subjects who experience any clinically significant AE will remain under medical supervision until the Investigator or the Sponsor's Medical Monitor deems the AE to be resolved, stabilized, or no longer serious enough to warrant follow-up.

## 3.6.5. Pregnancy reporting

Prior to study enrollment, females of childbearing potential must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. The signed Informed Consent Form must document this discussion.

A UPT will be performed on all females of childbearing potential at Day 1 (day of first patch application) and EOS. All women of childbearing potential will receive a UPT prior to the first study drug administration and the study drug must be withheld until the results of laboratory pregnancy testing are available. If pregnancy is confirmed, the subject must not receive any study drug and must not be enrolled in the study.

## 3.6.6. Expected Adverse Events

Any observed response in the patch test area that can be denoted using the irritation criteria summarized in Table 3 and Table 4 will not be considered an AE.

Tape related reactions will only be recorded as AEs when the subject is discontinued due to tape reaction around all sites. When 1 or 2 sites are experiencing severe tape related reactions, the application site will be stopped and the subject will continue on the study.

# 3.7. Instructions for Rapid Notification of Serious Adverse Events

#### 3.7.1. Contact person and number

Serious adverse events must be reported immediately (i.e., not later than 24 hours after first knowledge) by e-mail with the scanned TKL SAE report form to:



## 3.7.2. Reporting Responsibility

Any death, SAE, pregnancy, (see Section 3.6), or unusual frequency of AEs, must be reported immediately (i.e., not later than 24 hours after first learning of its occurrence) to the Sponsor's study manager by the Investigator, even if the event(s) appear to be unrelated to study treatment. Follow-up information about a previously reported SAE or pregnancy must also be reported to the Sponsor within 24 hours of receiving it. If the SAE or pregnancy has not been previously documented (i.e., is a new occurrence) and it is thought to be related to the investigational product (or therapy), the Sponsor may contact the Investigator to obtain further information. If warranted, an investigator alert may be issued, to inform all Investigators involved in any study with the same product (or therapy) that this SAE or pregnancy has been reported.

The IRB should also be notified of SAEs or pregnancies and of any follow-up information in writing, as is practical, and depending on local regulations.

## 3.7.3. Reporting procedures

For each SAE, the Investigator will complete a SAE Report Form in English and assess the relationship of each SAE to study treatment. The completed form(s) should be sent by e-mail to the Sponsor within 24 hours of first knowledge of the SAE (as outlined in Section 3.7.1 and Section 3.7.2). The initial SAE should be reported immediately, even if only preliminary information is available. Follow-up information should be sent by the same Investigator, restating the date of the original report. Either a new SAE form is sent (stating that it is a follow-up), or the original one is resent (with the new information highlighted and a new date provided). The follow-up should describe whether the event has resolved or continues, if and how it was treated, whether the blind was broken or not, and whether the patient continued or discontinued study participation. The form confirmation will be retained.

Pregnancy follow-up (as outlined in Section 3.6.5) should be reported to the IRB within 24 hours of first knowledge on a Pregnancy Report Form. Follow up will describe the outcome of the pregnancy, including any voluntary or spontaneous termination, details of the birth, and the presence or absence of any congenital abnormalities or birth defects.

# 3.8. Appropriateness of Safety Measurements

The safety assessments in the study are standard safety measures in clinical trials.

## 4. STATISTICAL METHODS

# 4.1. General Considerations for Data Analysis

The focus of the statistical analysis will be the comparison with controls of the photoallergic response to the study products. The diagnosis of photosensitization response will be made by the Investigator based on review of the observed skin responses after Challenge.

The mean score by subject and treatment, including all scores assigned during Induction, will be analyzed in the analysis of variance with factors subject and treatment. All pairwise treatment comparisons will be performed.

All statistical processing will be performed using the SAS® system (version 9.2 or higher). No interim or subgroup analyses are planned.

# 4.2. Sample Size and Power Considerations

The sample size of 50 evaluable subjects conforms to industry and regulatory standards for determination of irritation/sensitization when topical application to skin is followed by light exposure.

# 4.3. Subject Populations for Analysis

All subjects who receive treatment will be evaluable for AEs. The evaluation of photosensitization will be based on all subjects who complete the Challenge Phase of the study. Subjects who completed Challenge are those who have received at least 6 applications/irradiation of study products, and at least 11 subsequent evaluations during Induction, completed the Rest Phase and have received one application of study products at Challenge, subsequent irradiation and at least 4 evaluations (3 post-irradiation evaluations) for that product. The analysis of local tolerability (photo irritation) will be based off all subjects who complete the Induction Phase of the study. Subjects who completed Induction are those who have received at least 6 applications/irradiation of study products, and at least 11 subsequent evaluations during Induction.

## 4.3.1. Background and Demographic Characteristics

Descriptive statistics will be used to summarize demographic characteristics (age, gender, Fitzpatrick skin type, and race) and background characteristics for the randomized subject population. Past/coexistent medical history information for all randomized subjects will be presented in a by-subject listing.

## 4.3.2. Study Product/Visit Compliance

Descriptive statistics will be used to summarize study product compliance for the randomized subject population.

## 4.4. Prior and Concomitant Medications

Prior and concomitant medication information for all randomized subjects will be presented in a by-subject listing.

# 4.5. Efficacy Evaluation

This section is not applicable to this study.

# 4.6. Safety Evaluation

#### 4.6.1. Assessment of Responses

All assigned scores during Induction and Challenge will be summarized by frequency counts by time point and treatment. The incidence of reactions will be summarized by frequency counts for each treatment. The mean score by subject and treatment, including all scores assigned during Induction, will be analyzed using Fisher's least significant differences in the analysis of variance (ANOVA) with factors subject and treatment. All pairwise comparisons will be performed: CCP-020 (Diacerein 1%) topical ointment on both the irradiated and non-irradiated sides, and vehicle ointment on both the irradiated and non-irradiated sides.

## 4.6.2. Photosensitivity

The determination of dermal photosensitization potential will be made by the Investigator based on specific scoring criteria derived from observations in the Challenge Phase of the study and confirmed in the Rechallenge Phase, if necessary. The incidence of photosensitization reactions will be summarized by frequency counts for each treatment. If photosensitization occurs, the 95% confidence interval for the proportion of subjects with photosensitization for each product will be calculated. Photosensitivity will not be determined by statistical methods.

#### 4.6.3. Adverse Events

Adverse events will be summarized as an overall incidence of at least one event, incidence within body systems only, incidence by body system and preferred term, and by highest severity. Each subject will contribute only once (e.g., the first occurrence) to each of the rates, regardless of the number of occurrences (events) the subject experiences.

Treatment-emergent AEs will be summarized and tabulated by the system organ class and preferred term, by severity (mild, moderate, severe) and by relationship to study product (not related, unlikely, possible, probable, and definite).

Treatment-emergent will be defined as any AE with an onset date on or after the first study product administration date. Any event with a missing onset date will be included as a treatment-emergent AE.

Deaths and SAEs will be listed by subject.

# 4.7. Other topics

There are no other topics being evaluated.


# 4.8. Interim analyses

No interim analyses are anticipated.

# 4.9. Special Methods

This section is not applicable for this protocol.

## 5. ADMINISTRATIVE PROCEDURES

## 5.1. Ethics and Good Clinical Practice

This study must be carried out in compliance with the protocol and in accordance with TKL Research, Inc.'s standard operating procedures. These are designed to ensure adherence to Good Clinical Practices guidelines, as described in:

- ICH Harmonized Tripartite Guidelines for Good Clinical Practice 1996. Directive 91/507/EEC, The Rules Governing Medicinal Products in the European Community.
- US 21 Code of Federal Regulations dealing with clinical studies (including parts 50 and 56 concerning informed consent and IRB/IEC/EEC regulations).
- Declaration of Helsinki, concerning medical research in humans (Recommendations Guiding Physicians in Biomedical Research Involving Human Subjects, Helsinki 1964 and amendments).

The PI agrees, when signing the protocol, to adhere to the instructions and procedures described in it and thereby to adhere to the principles of GCP that it conforms to.

## 5.2. Institutional Review Board

Before implementing this study, the protocol, the ICF and other information to subjects, must be reviewed by a properly constituted IRB. A signed and dated statement that the protocol and informed consent have been approved by the IRB must be given to Sponsor before study initiation. This committee must also approve any amendments to the protocol, other than administrative ones, and a signed and dated statement of approval must be sent to the Sponsor prior to initiation of the amendment procedures. The name and occupation of the chairman and the members of the IRB must also be supplied to Sponsor.

## 5.3. Informed consent

The Investigator must explain to each subject (or legally authorized representative) the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits involved, and any discomfort it may entail. Each subject must be informed that participation in the study is voluntary, that he/she may withdraw from the study at any time, and that withdrawal of consent will not affect his/her subsequent medical treatment or relationship with the treating physician.

This informed consent should be given by means of a standard written statement, written in non-technical language. The subject should read and consider the statement before signing and dating it, and he/she should be given a copy of the signed document. No subject can enter the study before informed consent has been obtained from him/her, or his/her legally authorized representative.

The ICF is considered to be part of the protocol, and must be submitted by the PI with it for IRB approval. Any changes to the proposed ICF suggested by the PI must be agreed to by Castle

Creek Pharmaceuticals, LLC before submission to the IRB and a copy of the approved version must be provided to Castle Creek Pharmaceuticals, LLC after IRB approval.

## 5.4. Declaration of Helsinki

The PI must conduct the study in accordance with the laws and regulations of the country in which the study is conducted, as outlined in the Declaration of Helsinki.

# 5.5. Changes in Planned Study Conduct

#### 5.5.1. Protocol amendments

With the exception of changes in the visit schedule and/or administrative changes, any changes or additions to this clinical study protocol require a written protocol amendment that must be approved by Castle Creek Pharmaceuticals, LLC and the PI before implementation. Amendments significantly affecting the safety of subjects, the scope of the investigation or the scientific quality of the study, require additional approval by the appropriate IRB. A copy of the written approval of the IRB, which becomes part of the protocol, must be given to Castle Creek Pharmaceuticals, LLC. Examples of amendments requiring such approval are:

- 1. an increase in study product dosage or duration of product exposure of subjects,
- 2. a significant change in the study design (e.g., addition or deletion of a control group),
- 3. an increase in the number of invasive procedures to which subjects are exposed, and
- 4. addition or deletion of a test procedure for safety monitoring.

These requirements for approval should in no way prevent any immediate action from being taken by the Investigator or the Sponsor in the interests of preserving the safety of all subjects included in the study. If an immediate change to the protocol is felt to be necessary by the Investigator and is implemented by him/her for safety reasons the study Sponsor should be notified and the IRB should be informed within 10 working days.

Amendments affecting only administrative aspects of the study do not require formal protocol amendments or IRB approval, but the IRB must be kept informed of such administrative changes. Examples of administrative changes not requiring formal protocol amendments and IRB approval that can be treated as administrative amendments include:

- 1. changes in the staff used to monitor studies, and
- 2. minor changes in the packaging or labeling of the study product.

## 5.5.2. Other changes in study conduct

Deviations from the planned study conduct are not permitted; any unforeseen changes in study conduct must be reported to the Sponsor and noted in the final clinical study report.

## **5.5.3.** Termination or suspension of study

Both the Sponsor and the PI reserve the right to terminate or suspend the study at any time. If study termination is necessary, the procedures will be arranged on an individual study basis after

review and consultation by both parties. It is the responsibility of the PI to notify the IRB of the termination/suspension and the reason(s). In terminating the study, the Sponsor and the PI will ensure that adequate consideration is given to the protection of the subjects' interests.

## 5.6. Data handling and record keeping

#### 5.6.1. Recording of data

Case report forms will be designed to identify each subject by subject entry number and, where appropriate, subject's initials, the product being evaluated, and the results observed. All entries to the CRFs must be made as instructed by the study Sponsor at study initiation. Data on subjects collected on CRFs during the study will be documented in an anonymous fashion, and the subject will only be identified by the subject number, and by his/her initials, if also required. If, as an exception, it is necessary for safety or regulatory reasons to identify the subject, both the study Sponsor and the PI are bound to keep this information confidential.

The PI must sign the designated page(s) of the CRFs, thereby stating that he/she takes responsibility for the accuracy of the data in the entire case record book. All records will be kept in conformance to applicable national laws and regulations.

The original signed ICF will be attached to each subject's file. When the study treatment is completed, the ICF will be kept in the appropriate file folder; otherwise a note indicating where the records can be located will be made.

#### **5.6.2.** Retention of documents

Storage is maintained for 5 years or until the Sponsor advises to release the archives at either the TKL facility at One Promenade Blvd. Suite 1101/1201, Fair Lawn, NJ 07410 in a secured room accessible only to TKL employees, or at an offsite location that provides a secure environment with burglar/fire alarm systems, camera detection, and controlled temperature and humidity. Originals or copies of the CRFs, source documents, correspondence, IRB documents, study reports, etc. will be available for the Sponsor's review on the premises of TKL or at a secure location off-site. All database management activities can be found in the data management plan (DMP).

# 5.7. Product handling and accountability

All product supplies are to be used only for this clinical study and not for any other purpose. Study product supplies must be kept in an appropriate, secure area (e.g., locked cabinet) and stored according to the conditions specified on the product labels.

The PI or a designee must maintain a full record of the shipment and application of study product in a product accountability ledger. This log must be kept current and should contain the following information:

- identification of the subject to whom the study product was dispensed,
- date(s) of the study product dispensed to the subject, and
- initials of the study site representative(s) dispensing study product.

The inventory must be available for inspection by the study monitor. A product-inventory and storage-facility inspection will be conducted at appropriate time intervals throughout the clinical investigation, depending on enrollment and the length of the study. Any discrepancy and/or deficiency must be accounted for by the PI or his/her designee.

The PI must not destroy any product labels, or any partly used or unused product supply. At the conclusion of the study and, as appropriate, during the course of the study, all study product supplies, including partially used or empty containers, must be returned according to the designation of the Sponsor. Any missing supplies will be indicated on the inventory; the original inventory list will be retained in the PI's records for this clinical study.

# 5.8. Quality control and quality assurance

## **5.8.1.** Monitoring procedures

During the study, the Sponsor may visit the site regularly to check the completeness of subject records, the accuracy of entries on the CRFs, the adherence to the protocol and to ICH-GCP guidelines, the progress of enrollment, and also to ensure that study product is being stored, dispensed and accounted for according to specifications. Key investigative personnel will be available to assist the field monitor during these visits.

The data required by the protocol must be recorded on the appropriate CRFs. The CRFs and any source documents will be available to the study monitor who will perform a 100% data check (comparison of the data recorded in the CRF with those in the source documents). The CRFs and source data will also be available for an audit by the Sponsor or the FDA at any time.

The Investigator will give the monitor access to relevant clinical records, to confirm their consistency with the CRF entries. No information in these records about the identity of the subjects will leave the study center. Additional checks of the consistency of the source data with the CRFs are performed according to the study-specific monitoring plan.

## **5.8.2.** Auditing procedures

In addition to the routine monitoring procedures, a study center may be audited in depth for study quality assurance by the Sponsor, an external auditor on behalf of the Sponsor, and/or by regulatory authorities. This audit may include a review of all source documents, drug records, and original CRFs the study site used in this study. Patient confidentiality will be maintained at all times and consent for this will be obtained before entry of the patient into the clinical study (see Section 5.3). If an inspection is requested by a regulatory authority, the PI must immediately inform the study Sponsor that this request has been made.

# 5.9. Confidentiality and publication policies

#### 5.9.1. Disclosure and confidentiality

By signing the protocol, the PI agrees to keep all information provided by the Sponsor in strict confidence and to request similar confidentiality from his/her staff and the IRB. Study documents provided by the Sponsor (protocols, IBs, CRFs and other material) will be stored appropriately to ensure their confidentiality. The information provided by the Sponsor to the PI


may not be disclosed to others without direct written authorization from the Sponsor, except to the extent necessary to obtain informed consent from subjects who wish to participate in the study.

## 5.9.2. Communication and publication of results

Any formal presentation or publication of data from this study will be considered as a joint publication by the Investigator(s) and appropriate Sponsor personnel. Authorship will be determined by mutual agreement.

Castle Creek Pharmaceuticals, LLC must receive copies of any intended communication in advance of publication (at least 15 working days for an abstract or oral presentation and 45 working days for a journal submission). The Sponsor will review the communications for accuracy (thus avoiding potential discrepancies with submissions to health authorities), verify that confidential information is not being inadvertently divulged and provide any relevant supplementary information.

## 6. REFERENCES

- 1. Investigator's Brochure. CCP-020 (Diacerein 1%) Topical Ointment. Castle Creek Pharmaceuticals, LLC. Version Number 1.0. 04 November 2016.
- 2. Berger DS. Specification and design of solar ultraviolet simulators. Journal of Investigational Dermatology. 1969; 53:192-199.
- 3. Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch.Dermatol. 1988; 124: 869-871.
- 4. Sachdeva S. Fitzpatrick skin typing: Applications in dermatology. Indian J Dermatol Venereol Leprol 2009; 75:93-6



,

